CLINICAL TRIAL: NCT06758323
Title: Effect of Beetroot Juice Supplements with Caffeine Co-ingestion on Lower-limb Strength in Females
Brief Title: Acute Effects of Beetroot Juice and Caffeine Co-ingestion on Lower-limb Strength and Muscular Endurance in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Manuel Jurado Castro (Other)
Responsible Party: Sponsor-Investigator, Jose Manuel Jurado Castro, Principal Investigator, Maimónides Biomedical Research Institute of Córdoba
Organization: Maimónides Biomedical Research Institute of Córdoba (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IMIBIC_BRJ_CAF
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Beetroot Juice; Caffeine; Placebo; Beetroot Juice with Caffeine Co-ingestion
Keywords: beetroot juice; nitrate; caffeine; resistance training; dietary supplement; female
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Double-Blind Crossover Randomized Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- COM (Experimental): Beetroot juice combined with caffeine
  Interventions: Dietary Supplement: Beetroot juice combined with caffeine (COM)
- CAF (Active Comparator): Beetroot juice placebo with caffeine
  Interventions: Dietary Supplement: Beetroot juice placebo with caffeine (CAF)
- BRJ (Active Comparator): Beetroot juice with caffeine placebo
  Interventions: Dietary Supplement: Beetroot juice with caffeine placebo (BRJ)
- PLA (Placebo Comparator): Beetroot juice placebo with caffeine placebo
  Interventions: Other: Beetroot placebo with caffeine placebo (PLA)

INTERVENTIONS:
Dietary Supplement: Beetroot juice combined with caffeine (COM) — * 70 mL of beetroot juice (400 mg NO3-, BEET It Sport; James White Drinks Ltd) 120 minutes before experimental session
  * 200 mg caffeine capsule from the IO.GENIX Nutrition brand (Toledo, Spain) 60 minutes before experimental session
  Arms: COM
Dietary Supplement: Beetroot juice placebo with caffeine (CAF) — - 70 mL of a blackcurrant beverage, which depletes NO3- (Capri-Sun) 120 minutes before experimental session - 200 mg caffeine capsule from the IO.GENIX Nutrition brand (Toledo, Spain) 60 minutes before experimental session
  Arms: CAF
Dietary Supplement: Beetroot juice with caffeine placebo (BRJ) — - 70 mL of beetroot juice (400 mg NO3-, BEET It Sport; James White Drinks Ltd) 120 minutes before experimental session - Multivitamin capsule from NaturrTierra (Leganés, Spain) 60 minutes before experimental session
  Arms: BRJ
Other: Beetroot placebo with caffeine placebo (PLA) — - 70 mL of a blackcurrant beverage, which depletes NO3- (Capri-Sun) 120 minutes before experimental session - Multivitamin capsule from NaturrTierra (Leganés, Spain) 60 minutes before experimental session
  Arms: PLA

SUMMARY:
The aim of this study is to evaluate the acute effects of beetroot juice and caffeine, consumed individually or in combination, on lower-limb strength and muscular endurance in physically active women. The main questions it aims to answer are:

* Does the co-ingestion of beetroot juice and caffeine enhance lower-limb strength and muscular endurance more than either substance alone or a placebo?
* How do the acute effects of beetroot juice interact with caffeine on physical performance?

The study was conducted using a randomized, crossover design to evaluate the following four conditions:

Beetroot juice with placebo Caffeine with placebo Beetroot juice with caffeine Placebo only

Each participant completed all conditions, with a sufficient washout period between sessions to eliminate potential carryover effects. This design allowed for a direct comparison of the acute effects of each supplementation strategy on lower-limb strength and muscular endurance.

Participant Protocol

Participants consumed their assigned supplement on a single testing day for each condition. After supplementation, they performed standardized tests to measure lower-limb strength and muscular endurance. Progress was monitored, and data from all conditions were collected to assess the acute effects of each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Minimal experience of six months of strength training
* Be familiarized with the exercise test: counter movement jump (CMJ), barbell back squats, leg press and knee extension.

Exclusion Criteria:

* Supplementation consumption
* Sports injuries

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Change of height reached in jump | Visit 1 (Day 1), Visit 2 (Day 5), Visit 3 (Day 9), Visit 4 (Day 13)
  Evaluated through Countermovement jump test with a recovery period of 45 seconds between jumps. The height reached was recorded in centimeters.

SECONDARY OUTCOMES:
Movement velocity | Visit 1 (Day 1), Visit 2 (Day 5), Visit 3 (Day 9), Visit 4 (Day 13)
  The velocity was recorded in meters per second (m/s) during two repetitions of the back squat, evaluated at 50% and 75% of the repetition maximum (RM).
Muscular endurance test | Visit 1 (Day 1), Visit 2 (Day 5), Visit 3 (Day 9), Visit 4 (Day 13)
  The test consists of three exercises: back squat, leg press and leg extension. Three series will be performed until concentric failure at 75% RM, three minutes of rest between each series (3 series). The number of repetitions was recorded.
Rating of perceived exertion (RPE). | Visit 1 (Day 1), Visit 2 (Day 5), Visit 3 (Day 9), Visit 4 (Day 13)
  Immediately at the end of the muscular endurance test, participants will be instructed to report their RPE using a scale 1-10 (worse to better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Edificio IMIBIC Avda Menéndez Pidal s/n, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No